CLINICAL TRIAL: NCT01890915
Title: Core Temperature During Heat Exposure in Persons With Tetraplegia
Brief Title: Body Temperature in Persons With Tetraplegia When Exposed to Heat
Status: Completed | Type: Observational
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, John Handrakis, PT, DPT, EdD, Research Health Science Specialist, James J. Peters Veterans Affairs Medical Center
Other Study IDs: HAN-12-04
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; Body temperature; Executive function; Sweat
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tetraplegia: Persons with spinal cord injury, level of injury C4-T1, American Spinal Injury Association (ASIA) impairment levels A-B and duration of injury greater than 1 year. Ages 18-65 years old.
  Interventions: Other: Heat Exposure
- Control: Age and gender-matched able-bodied controls. Ages 18-65 years old.
  Interventions: Other: Heat Exposure

INTERVENTIONS:
Other: Heat Exposure — Heat exposure of 95 degrees F for up to 2 hours.
  Other Names: 95 degrees F for up to 2 hours.

SUMMARY:
The deleterious effects of hyperthermia are well appreciated in able-bodied persons. However, the consequences of impaired regulation of normal body temperature on cognitive performance of persons with tetraplegia is not known. This study will provide the preliminary findings necessary for future work to design and explore physical and medical interventions to improve temperature regulation in those with tetraplegia with the goal of improved clinical care, health, and quality of life.

The proposed study consists of 1 visit during which 20 subjects (10 with tetraplegia, 10 controls) will be exposed to 81°F for 40 minutes and then 95° F for up to 2 hours. Physiological as well as psychological processes will be monitored in all subjects during the study for safety and to determine differences in responses to exposure to hot ambient temperatures

DETAILED DESCRIPTION:
After a cervical spinal cord injury (SCI) the motor, sensory and autonomic deficits cause, among other detriments, a blunted ability to maintain a constant core temperature. Impaired thermoregulation leaves persons with tetraplegia more susceptible to hyperthermia than able-bodied persons (AB). There has been a paucity of work addressing the thermoregulatory responses of persons with SCI to hot ambient temperatures, and even less study addressing the effect of these temperatures on cognitive performance. The goals of this pilot study are: to improve our understanding of the thermoregulatory mechanisms of individuals with tetraplegia when exposed to heat and to determine the effect of impaired thermoregulatory mechanisms on cognitive performance during exposure to 35°C for up to 2 hours. In order to address our goals we have designed a study methodology which consists of comparing the physiological and psychological responses of the two study groups (tetraplegia versus AB controls) from thermoneutral (27°C) to hot (35°C) environments.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 65 years of age;
2. Duration of injury ≥ 1 year;
3. Level of SCI C4-T1;
4. Euhydration (Subjects will be instructed to avoid caffeine and alcohol, maintain normal salt and water intake, and avoid strenuous exercise for 24 hours prior to study); and
5. Age (± 5 years) and gender matched AB control group.

Exclusion Criteria:

1. Known heart and/or blood vessel disease;
2. High blood pressure;
3. Kidney disease;
4. Diabetes mellitus;
5. Acute illness or infection;
6. Dehydration;
7. Pregnant women;
8. Untreated thyroid disease, and
9. Broken, inflamed, or otherwise fragile skin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 subjects with tetraplegia (SCI, C4-T1), ages 18-65 years old and 10 age- and gender-matched, able-bodied controls will be accepted for participation.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Handrakis, PT, DPT, EdD, Principal Investigator — Center of Excellence for the Medical Consequences of SCI, James J Peters VAMC
Locations (1):
- Center of Excellence for the Medical Consequences of SCI, James J Peters VAMC, The Bronx, New York, United States

REFERENCES:
- [Derived] Kumar NS, Bart J, Barton C, Graham ML, Leung PP, Tittley TD, Lee I, Bang C, Bauman WA, Handrakis JP. Core Temperature Lability Predicts Sympathetic Interruption and Cognitive Performance during Heat Exposure in Persons with Spinal Cord Injuries. J Neurotrauma. 2021 Aug 1;38(15):2141-2150. doi: 10.1089/neu.2020.7598. Epub 2021 May 26. PMID 33882698
- [Derived] Handrakis JP, Ni Guan Z, Nulty JW, Tascione O, Rosado-Rivera D, White D, Bang C, Spungen AM, Bauman WA. Effect of Heat Exposure on Cognition in Persons with Tetraplegia. J Neurotrauma. 2017 Dec 15;34(24):3372-3380. doi: 10.1089/neu.2016.4850. Epub 2017 Aug 16. PMID 28462685

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tetraplegia | Control
Started | 11 | 10
Completed | 8 | 9
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Equipment Malfunction | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Tetraplegia: Persons with spinal cord injury, level of injury C4-T1, ASIA levels A-B and duration of injury greater than 1 year. Ages 18-65 years old.
  Heat Exposure: Heat exposure of 95 degrees F for up to 2 hours.
- Total: Total of all reporting groups
Arm/Group | Tetraplegia | Control | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Core Body Temperature
Description: To determine the change in core body temperature in the seated position from 79 degrees F for 30 minutes to 95 degrees F for up to 2 hours. Hypotheses: Persons with tetraplegia will have a greater increase in core body temperature than able-bodied (AB) control subjects. Core body temperature in AB persons will be maintained.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Tetraplegia | Control
Number analyzed (Participants) | 8 | 9
Percent Change | 2.04 (0.49) | -0.05 (0.61)
Statistical Analysis 1: Comparison: Tetraplegia vs Control; Due to impaired thermoregulatory mechanisms secondary to spinal cord injury, subjects with tetraplegia were hypothesized to have a significant rise in core temperature after exposure to warm ambient temperatures, while control subjects were hypothesized to maintain constant core temperature. Percent change in core temperature of subjects in each group were compared to determine if they were significantly different from baseline to warm exposure; Test type: Superiority or Other; p = 0.0001, ANOVA

2. Secondary Outcome: Cognitive Performance - Stroop Interference T-Scores
Description: To determine the change in cognitive performance as measured by the Stroop Color and Word Interference T-Scores, measured after 30 min at 79 degrees F and after up to 2 hours at 95 degrees F. Interference T-Scores are derived from the difference between the raw Color-Word score and the projected Color-Word score (which is, in turn, based on the raw scores obtained in the Word and Color portions of the Test). Lower scores indicate poorer performance, and a positive percent change in T-scores indicates improved performance. Hypothesis: Persons with tetraplegia compared with AB will have a greater change in cognitive performance from baseline (79 degrees) to warm exposure (95 degrees).
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tetraplegia | Control
Number analyzed (Participants) | 8 | 9
Percent change | 8.3 (5.9) | 0.3 (6.6)
Statistical Analysis 1: Comparison: Tetraplegia vs Control; We hypothesized that subjects with tetraplegia would demonstrate a change in cognitive performance after heat exposure if they had demonstrated a significant increase in core body temperature - as was hypothesized in our primary hypothesis. Cognitive performance was measured, in part, by Interference T-scores derived from the Stroop Color and Word Test; Test type: Superiority or Other; p = 0.006, ANOVA

3. Other Pre Specified Outcome: Sweat Rate
Description: To determine the change in sweat rate using QSweat methodology (WR TestWorks) from 30 minutes at 79 degrees F compared to after up to 2 hours at 95 degrees F. Sweat collection capsules will be placed on the left lateral anterior shoulder, volar aspect of the distal forearm, proximal anterior thigh, and mid-lateral calf (dermatomes C5, T1, L3, L5) for measurement of sweat rate. Hypothesis: Persons with tetraplegia compared with AB will have less of a percent change in average sweat rate after heat exposure.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tetraplegia | Control
Number analyzed (Participants) | 8 | 9
Percent change | 51.4 (12.6) | 1030.2 (654.9)
Statistical Analysis 1: Comparison: Tetraplegia vs Control; Due to impaired thermoregulatory mechanisms, subjects with tetraplegia were hypothesized to have diminished increases in sweat rate in comparison to controls after heat exposure; Test type: Superiority or Other; p = 0.015, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were reported within five business days to the VA's Institutional Review Board (IRB) via an Adverse Event form and were also included on the Adverse Events log on the annual continuing review application in accordance with VA IRB policy.
Description: Adverse event data were collected throughout the entire course of the study, i.e. from 2012 to 2015.
Arm/Group | Tetraplegia | Control
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tetraplegia (N=11) | Control (N=10)
Autonomic dysreflexia (Nervous system disorders) | 1 (1) | 0 (0) — Subject experienced autonomic dysreflexia (AD), presenting with high blood pressure, flushing, and diaphoresis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes